CLINICAL TRIAL: NCT02057432
Title: A Pilot Study to Evaluate Image-guided Breast Conserving Surgery in the Advanced Multimodality Image Guided Operating Suite (AMIGO)
Brief Title: Image-guided Breast Surgery in the Advanced Multimodality Image Guided Operating Suite (AMIGO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Mehra Golshan, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 11-454
Record Dates: First submitted 2014-01-03; First posted 2014-02-07 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Stage I Breast Carcinoma; Stage II Breast Carcinoma
Keywords: I-II Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intra-operative MRI (Experimental): Images will be obtained both before and after intravenous bolus injection with subsequent dynamic imaging. Dynamic contrast enhancement maps will be created for evaluation of residual tumor. Images will be reformatted into three orthogonal planes as well as into a 3D model for surgical orientation. All imaging protocols using contrast, contrast enhancement maps and reformatting, as described above, which will be applied to the intra-operative MRI performed in the AMIGO suite are consistent with the standard MRI breast imaging at Brigham and Women's Hospital.
  Interventions: Device: intra-operative MRI

INTERVENTIONS:
Device: intra-operative MRI — Patients will undergo an MRI during surgery.

SUMMARY:
This research study is a pilot study designed to evaluate magnetic resonance imaging-guided therapy (MRT) as a possible treatment for breast cancer. In this pilot study, the investigators are studying if it is possible to use intra-operative MRI to guide surgery. The therapy takes place in the Advanced Multimodality Image Guided Operating (AMIGO) suite at Brigham and Women's Hospital.

The purpose of this study is to investigate if it is possible to perform the breast conserving surgery with the help of intra-operative magnetic resonance imaging in the advanced multimodality image guided operating suite. It is hoped that intra operative MRI may improve the surgeon's ability to know the exact margins of tumor. Currently, approximately 40% of women need to come back to the operating room and have the margins of the cancer re-excised.

DETAILED DESCRIPTION:
The treatment being studied consists of standard lumpectomy and sentinel node biopsy if indicated, or standard axillary dissection if clinically indicated. The study includes the additional use of MRI to guide the removal of the cancer. The MRI uses powerful magnets linked to a computer to create detailed pictures of the breast. The purpose of the current study is to find out whether performing the intra-operative MRI is possible, safe and practical. As part of the study the participant will need to have tests to show that they are eligible to participate in the research study.If the participant does not meet the eligibility criteria, they will not be able to participate in this research study.

Surgery Day

* Wire localization with ultrasound, Mammogram or MRI in the non-palpable tumor is placed in the participant's breast. The presence of the wire in the tumor will then help guide the surgeon to the location of the tumor.
* The sentinel node biopsy or axillary dissection will be performed if indicated.
* Then the lumpectomy will be performed.
* The participant will undergo an intra-operative MRI scan in the AMIGO.

  ---If the MRI images indicate there may be tumor behind, more tissue will be removed from the respective margins. No additional MRIs will be performed.
* Most of these operations are outpatient. However, the need to stay overnight may occur if the recovery from anesthesia is slow or if the participant underwent an axillary dissection.

Within six weeks after patient surgery. The participant will have the following procedures:

* History and physical exam
* Wound check
* The participant will also be informed of the final pathology, including margin status.The remainder of follow up will be as per standard of care after breast conserving surgery for breast cancer. The participant will be assessed by physical exam for possible complications and local recurrence. These visits will likely overlap with established oncology care team follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a pre-operative standard mammogram with or without ultrasound. These may be performed at outside institutions.
* Participants must have biopsy confirmed invasive breast carcinoma. If biopsy was done at an outside hospital, pathology will be reviewed at BWH/DFCI.
* Stage: Clinical Staging must be Stage I or II as outlined by the AJCC 7th edition. Pre-operative diagnosis of positive axillary nodes necessitating axillary dissection at the time of lumpectomy does not disqualify a patient.
* Pre-operative sentinel node biopsy also does not disqualify the patient.
* Participants must be candidates for definitive local therapy with breast conserving therapy (this takes into account tumor to breast size ratio appropriate for BCS, and the ability to undergo standard radiation therapy post-operatively).
* Participants must have measurable disease, defined as one lesion that can be accurately measured by MRI. (More than one lesion will be an exclusion criteria for BCS; lesions not identified by MRI will also be an exclusion criteria).
* Age ≥ 18 years and < 75.
* Completion of the magnetic resonance (MR) procedure screening form and clearance by the MR technologist that the patient does not have a pacemaker, brain aneurysm clip, inner ear implant, neurostimulator or metal fragments in the eye.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Participants with a known BRCA 1 or 2 mutation.
* Participants with known Li-Fraumeni or Cowden's Disease.
* Participants with prior mantle radiation.
* Participants with locally advanced breast cancer such as inflammatory breast cancer or cancer grossly involving skin.
* Participants who are pregnant.
* Participants who enroll in a preoperative therapy trial or who have been treated with neoadjuvant chemotherapy. The neoadjuvant chemotherapy can result in complete pathologic response, resulting in no signal on MRI.
* Participants with known, active collagen vascular disease.
* Participants who undergo breast surgery at an outside institution.
* Participants with prior history of breast carcinoma.
* Patients who have implants or any type of breast reconstruction.
* Patients who have biopsy confirmed multi-centric disease.
* Participants who have documented contra-indications for MRI.
* Participants who have documented allergic reaction to IV MRI contrast agent, or have a contraindication to the administration of IV contrast such as renal failure.
* Patients with diabetes will be excluded because of a higher risk to incur renal damage from the IV contrast.
* Participants who exceed the weight limit for the surgical table at AMIGO, 350 lbs or who will not fit into the 70 cm diameter bore of the MRI scanner at AMIGO or the 60 cm diameter bore of the pre-procedure imaging MRI scanner.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To demonstrate feasibility of using the intra-operative MRI for breast conserving surgery | 2 Years
  For the purpose of this pilot study, feasibility is defined as the ability to successfully complete the breast conserving operation in the
  AMIGO suite. Feasibility must entail the following:
  All necessary instruments for this operation are MRI compatible or are able to be used safely and then stored outside of the magnetic field when the intra-operative MRI is performed. The intra-operative MRI is performed without compromising the sterile operative field.

SECONDARY OUTCOMES:
Duration of the Lumpectomy and Imaging | 2 Years
  To measure duration of the lumpectomy portion of the procedure, the duration of the imaging portion of the procedure, and time under anesthesia.
Final Pathology Report and Intra-operative MRI Comparison | 2 Years
  The intra-operative MRI images will be compared to final pathology report which is the gold standard. This objective is for the purpose of collecting preliminary data for planning a future study which will be adequately powered to show the sensitivity and true positives of the intraoperative MRI.
Number of operations needed to obtain clear margins if clear margins were not obtained on initial operation. | 2 Years
  Number of operations needed to obtain clear margins if clear margins were not obtained on initial operation.
Volume of tissue removed on initial operation and on secondary operations if these were necessary. | 2 Years
  Volume of tissue removed on initial operation and on secondary operations if these were necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Mehra Golshan, MD, Principal Investigator — Dana Farber Cance Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No